CLINICAL TRIAL: NCT06589674
Title: Comparison of the Effectiveness of Pleth Variability Index and Diastolic Shock Index in Predicting Hypotension During Anesthesia Induction
Brief Title: Comparison of Pleth Variability Index vs. Diastolic Shock Index for Predicting Hypotension During Anesthesia Induction
Status: Completed | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Yuksek, Md, Kocaeli City Hospital
Other Study IDs: 2024-69
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia Induced Hypotension; Hypotension Drug-Induced
Keywords: Anesthesia Induction; Hypotension Prediction; Pleth Variability Index (PVI); Diastolic Shock Index (DSI); Hemodynamic Monitoring
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General Anesthesia Group: This group includes all study patients who underwent elective lumbar spine surgery under general anesthesia. In these patients, both PVI and DSI measurements will be performed before and during anesthesia induction.
  Interventions: Diagnostic Test: Pulse variability index measurement; Other: Diastolic shock index

INTERVENTIONS:
Diagnostic Test: Pulse variability index measurement — Peripheral perfusion index (PI) is an easy-to-implement and low-cost monitoring procedure obtained by interpreting non-invasive data obtained from pulse oximetry via plethysmography. It is a tool that allows interpretation of fluid status through changes in pulse oximetry waves caused by respiration. High perfusion indices are interpreted as low arterial tone. Changes in perfusion index are interpreted as indicators of vascular tone or fluid deficit problems in patients. The ratio of the highest and lowest PI values gives the Pleth Variability Index (PVI) (3,4). Hypotension can be predicted during anesthesia induction with PVI
  Other Names: PVI
Other: Diastolic shock index — The Diastolic Shock Index (DSI) is a hemodynamic parameter calculated by dividing the heart rate (HR) by the diastolic blood pressure (DBP). It reflects the balance between cardiac output and systemic vascular resistance, particularly in critically ill patients. A higher DSI can indicate impaired vascular resistance and may be useful for predicting the need for vasopressor support, especially in conditions like septic shock. However, its application in predicting hypotension during anesthesia induction is still under investigation.
  Other Names: DSI

SUMMARY:
This study aims to explore the frequent occurrence of hypotension during anesthesia induction due to anesthetic drugs or fasting. Predicting this condition is important for patient safety and anesthesia management. The study examines two indices: the Pleth Variability Index (PVI), derived from pulse oximeter readings, and the Diastolic Shock Index (DSI), calculated using heart rate and diastolic blood pressure. While PVI is a well-known method, DSI has been less explored in predicting anesthesia-related hypotension. The study aims to compare the effectiveness of these two indices in forecasting hypotension during anesthesia induction.

DETAILED DESCRIPTION:
Hypotension is frequently observed during anesthesia induction due to the effects of anesthetic drugs on hemodynamics and the requirement of a specific fasting period before surgery. Induction-related hypotension can lead to decreased tissue perfusion and, consequently, secondary organ damage. Predicting anesthesia-induced hypotension in advance contributes to better anesthesia management and patient safety (1). Induction-related hypotension is defined as arterial hypotension occurring within the first 20 minutes after anesthesia induction or until the start of the surgery. Arterial hypotension is identified when mean systolic arterial pressure (MAP) decrease > 20% or MAP <65 mmHg or when norepinephrine is administered at a dose >;6 mcg/min at least once during this period (2).

The peripheral perfusion index (PI) is a simple, cost-effective monitoring method derived from non-invasive plethysmographic data using pulse oximetry. It provides an assessment of fluid status based on respiratory changes in pulse oximeter waves, with higher PI values indicating lower arterial tone. Changes in PI are interpreted as signs of vascular tone or fluid deficit issues in patients. The ratio of the highest and lowest PI values yields the Pleth Variability Index (PVI) (3,4). PVI can be used to predict hypotension during anesthesia induction (5).

Cardiac output (CO) is calculated by multiplying systemic vascular resistance (SVR) and heart rate (HR). In septic and shock patients, CO may be low, often due to decreased SVR. The autonomic system tries to maintain CO by increasing HR in response to the reduced SVR (6). Systolic and diastolic shock indices are obtained by dividing the HR by systolic and diastolic blood pressures, respectively. The diastolic shock index has been evaluated in studies to predict vasopressor response in septic patients (7). A high shock index has been associated with early vasopressor initiation and better prognosis. However, no study has yet examined the predictive power of the diastolic shock index, which is related to sympathetic response and systemic vascular resistance, for hypotension following anesthesia induction.

Moreover, the diastolic shock index has not been compared with the more commonly used PVI in terms of their ability to predict hypotension. Therefore, our study aims to test the success of diastolic shock index and PVI measurements in predicting anesthesia-induced hypotension

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a preoperative fasting period of at least 6 hours
2. Patients scheduled for elective surgery under general anesthesia
3. Patients aged 18-65 with ASA classification I-III
4. Patients undergoing lumbar spinal surgery

Exclusion Criteria:

1. Patients who do not agree to participate in the study
2. Emergency surgeries
3. Patients who will undergo surgery under spinal anesthesia
4. Patients diagnosed with autonomic neuropathy
5. Patients undergoing surgery with inotropic support

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo elective lumbar spine surgery in Kocaeli City Hospital operating rooms constitute the study universe.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Prediction of anesthesia-induced hypotension | First 20 minutes after induction of anesthesia
  Anesthesia-induced hypotension is a significant drop in blood pressure that occurs during the induction or maintenance of anesthesia.Arterial hypotension was defined as systolic blood pressure (SBP) ; 90 mmHg in at least one measurement during this period or norepinephrine administered at a dose of ;6 mcg/min at lea

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Yuksek, Associate Proffessor, Study Director — Kocaeli City Hospital; Ayse Sencan, Md, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing of patient data is prohibited by the institution and may be requested from the institution with appropriate request.

REFERENCES:
- [Background] Ospina-Tascon GA, Teboul JL, Hernandez G, Alvarez I, Sanchez-Ortiz AI, Calderon-Tapia LE, Manzano-Nunez R, Quinones E, Madrinan-Navia HJ, Ruiz JE, Aldana JL, Bakker J. Diastolic shock index and clinical outcomes in patients with septic shock. Ann Intensive Care. 2020 Apr 16;10(1):41. doi: 10.1186/s13613-020-00658-8. PMID 32296976
- [Background] Ospina-Tascon GA, Garcia-Gallardo G, Orozco N. Using the diastolic shock index to determine when to promptly administer vasopressors in patients with septic shock. Clin Exp Emerg Med. 2022 Dec;9(4):367-369. doi: 10.15441/ceem.22.401. Epub 2022 Dec 8. No abstract available. PMID 36480818
- [Background] Rasmy I, Mohamed H, Nabil N, Abdalah S, Hasanin A, Eladawy A, Ahmed M, Mukhtar A. Evaluation of Perfusion Index as a Predictor of Vasopressor Requirement in Patients with Severe Sepsis. Shock. 2015 Dec;44(6):554-9. doi: 10.1097/SHK.0000000000000481. PMID 26529657
- [Background] Coutrot M, Dudoignon E, Joachim J, Gayat E, Vallee F, Depret F. Perfusion index: Physical principles, physiological meanings and clinical implications in anaesthesia and critical care. Anaesth Crit Care Pain Med. 2021 Dec;40(6):100964. doi: 10.1016/j.accpm.2021.100964. Epub 2021 Oct 24. PMID 34687923
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Background] Kim YJ, Seo JH, Lee HC, Kim HS. Pleth variability index during preoxygenation could predict anesthesia-induced hypotension: A prospective, observational study. J Clin Anesth. 2023 Nov;90:111236. doi: 10.1016/j.jclinane.2023.111236. Epub 2023 Aug 26. PMID 37639751